CLINICAL TRIAL: NCT07042828
Title: An Open Label, Balanced, Randomized, Single Dose, Two Treatment, Two Sequence, Four Period, Full Replicate, Crossover, Oral Bioequivalence Study in Healthy, Adult, Human Subjects Under Fasting Condition
Brief Title: To Compare and Evaluate the Oral Bioavailability of Bilastine 20 mg Orally Dispersible Tablet With That of Bilaxten (Bilastine) 20 mg Orally Dispersible Tablet in Healthy, Adult, Human Subjects Under Fasting Conditions
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Humanis Saglık Anonim Sirketi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 25-VIN-0229
Record Dates: First submitted 2025-06-20; First posted 2025-06-29 (Actual); Last update posted 2025-06-29 (Actual); Status verified 2025-06

CONDITIONS: Allergic Rhino-Conjunctivitis; Urticaria
MeSH Terms: conditions — Urticaria | interventions — bilastine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bilastine oral dispersible tablets (Experimental): Bilastine 20 mg oral dispersible tablets
  Interventions: Drug: Bilastine oral dispersible tablets; Drug: Bilaxten oral dispersible tablets
- Bilaxten oral dispersible tablets (Active Comparator): Bilaxten 20 mg oral dispersible tablets
  Interventions: Drug: Bilastine oral dispersible tablets; Drug: Bilaxten oral dispersible tablets

INTERVENTIONS:
Drug: Bilastine oral dispersible tablets — Bilastine 20 mg oral dispersible tablets
Drug: Bilaxten oral dispersible tablets — Bilaxten 20 mg oral dispersible tablets

SUMMARY:
An open label, balanced, randomized single-dose, two-treatment, two sequence, four-period, Full Replicate, crossover oral bioequivalence study in healthy, adult, human subjects under fasting condition.

ELIGIBILITY:
Inclusion Criteria:

* Subjects aged between 18 and 45 years (both inclusive).
* Subjects' weight within normal range according to normal values for Body Mass Index (between 18.5 and 30.0 kg/m2) (both inclusive) with minimum of 45 kg weight.
* Subjects with normal health as determined by personal medical history, clinical examination and laboratory examinations within Predefined site Normal range [Annexure III (A)].
* Subjects having clinically acceptable 12-lead electrocardiogram (ECG).
* Subjects having clinically acceptable chest X-Ray (PA view), if taken.
* Subjects having negative urine screen for drugs of abuse (including amphetamines, barbiturates, benzodiazepines, marijuana, cocaine, and morphine).
* Subjects having negative urine alcohol test / breath alcohol test.
* Non-smoker.
* Subjects willing to adhere to the protocol requirements and to provide written informed consent.
* For male Subjects: Subjects willing to follow approved birth control methods (a double barrier method) for the duration of the study as judged by the investigator(s), such as (a double barrier method) condom with spermicide, Condom with diaphragm, or abstinence. Subjects willing to refrain from donating sperm during the study period
* For Female Subjects:

  * Female of child bearing potential practicing an acceptable method of birth control for the duration of the study as judged by the investigator(s), such as intrauterine device (IUD), abstinence, bilateral tubal ligation or double barrier contraception, i.e., condom + diaphragm, condom + spermicidal or foam
  * Postmenopausal for at least 1 year, or if less than 1 year, then following acceptable contraceptive measures as mentioned above
* Subjects having negative urine pregnancy test at screening and negative serum -hCG pregnancy test on admission day of period 01 (only for female subjects).

Exclusion Criteria:

* Hypersensitivity to Bilastine or related class of drugs or any of its excipients or heparin.
* History or presence of significant cardiovascular, pulmonary, hepatic, renal, gastrointestinal, endocrine, immunological, dermatological, neurological, urogenital or psychiatric disease or disorder.
* Any treatment which could bring about induction or inhibition of hepatic microsomal enzyme system within 30 days prior to admission in period 01.
* Presence of alcoholism or drug abuse.
* History or presence of asthma, urticaria or other significant allergic reactions.
* History or presence of significant gastric and/or duodenal ulceration.
* History or presence of significant thyroid disease, adrenal dysfunction, organic intracranial lesion such as pituitary tumor.
* History or presence of cancer or basal or squamous cell carcinoma.
* Difficulty with donating blood.
* Difficulty in swallowing solids dosage form like tablets or capsules.
* Use of any prescribed medication or OTC medication including vaccines, vitamins and herbal remedies during last 30 days prior to admission in period 01.
* Major illness within past 3 months.
* Volunteer who have donated blood (1 unit) or participation in a drug research study within past 90 days prior to the first dose of the study drug.
* Consumption of xanthine-containing products, tobacco containing products or alcohol or any alcohol containing products within 48.00 hours prior to admission in period 01.
* Consumption of grapefruit or grapefruit juice containing products within 72.00 hours prior to admission of period 01.
* Positive screening test for any one or more: HIV, Hepatitis B and Hepatitis C.
* History or presence of significant easy bruising or bleeding.
* History or presence of significant recent trauma.
* Subjects who have been on an abnormal diet (for whatever reason) during the four weeks preceding the study.
* Female subjects who are currently breast feeding.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 42 (Actual)
Dates: Start 2025-04-30 (Actual); Primary Completion 2025-06-16 (Actual); Study Completion 2025-06-19 (Actual)

PRIMARY OUTCOMES:
Peak Plasma Concentration (Cmax) | 24 hours
  90% confidence intervals for the geometric least squares mean ratio of (T/R) will be calculated and reported for Cmax
Area Under the Curve from time zero to time of last measurable concentration (AUC0-t) | 24 hours
  90% confidence intervals for the geometric least squares mean ratio of (T/R) will be calculated and reported for AUC0-t

SECONDARY OUTCOMES:
Area Under the Curve from time zero to time infinite (AUC0-∞) | 24 hours
  Description Statistics
Time to reach peak plasma concentration (Tmax) | 24 hours
  Description Statistics

CONTACTS AND LOCATIONS:
Locations (1):
- Veeda Clinical Research Ltd., Ahmedabad, Gujarat, India